CLINICAL TRIAL: NCT00006864
Title: Interleukin-2 In An Alternative Dose (The Iliad Trial): Treatment Of Patients With Metastatic Renal Cell Carcinoma With Low Dose Proleukin
Brief Title: Interleukin-2 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Chiron Corporation (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CHIR1899; CWRU-CHIR-1899; CHIR-MA-99-01; CWRU-010002; NCI-G00-1875
Record Dates: First submitted 2000-12-06; First posted 2003-06-02 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill kidney cancer cells.

PURPOSE: Phase IV trial to study the effectiveness of interleukin-2 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate, complete and partial response rates, and duration of response in patients with metastatic renal cell carcinoma treated with low-dose interleukin-2.
* Determine the overall survival, one-year progression-free survival, and two-year progression-free survival in patients treated with this regimen.
* Determine the incidence of adverse events in these patients.

OUTLINE: This is a multicenter study.

Patients receive low-dose interleukin-2 subcutaneously 5 days a week for 6 weeks. Courses repeat every 9 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 464 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic renal cell carcinoma

  * Clear cell
  * Papillary
  * Sarcomatoid
  * Mixed
* Measurable or evaluable disease
* Evidence of disease following surgical resection of metastases
* No CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10 g/dL
* WBC at least 4,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.8 mg/dL

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception (barrier plus 1 other method)
* Thyroid-stimulating hormone normal
* No known hypersensitivity or allergy to components of recombinant human interleukin-2
* No known autoimmune disease (e.g., Crohn's disease)
* No other concurrent medical condition that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior recombinant human interleukin-2
* No concurrent interferon alfa

Chemotherapy:

* No concurrent cytoxic chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy (e.g., medroxyprogesterone) other than estrogen replacement therapy
* No concurrent prophylactic glucocorticoids (replacement doses and topical use allowed)
* No concurrent systemic corticosteroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to index lesion
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Prior surgery for renal cell carcinoma allowed

Other:

* No prior systemic therapy for renal cell carcinoma
* At least 4 weeks since prior investigational drugs
* No other concurrent investigational drugs or participation in another clinical study
* No concurrent iodinated radiocontrast dye
* No concurrent drugs for another indication that has purported activity in treatment of neoplasia (e.g., thalidomide)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Connell, MD, PhD, Study Chair — University Hospitals Seidman Cancer Center
Locations (2):
- United States (2):
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - Ireland Cancer Center, Cleveland, Ohio